CLINICAL TRIAL: NCT03541304
Title: Efficacy and Toxicity of High Dose Radiotherapy Wich Concurrent Chemotherapy for the Treatment of Rectal Cancer
Brief Title: High Dose Radiotherapy for the Treatment of Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Professor, Sun Yat-sen University
Other Study IDs: 2018-FXY-079
Record Dates: First submitted 2018-05-18; First posted 2018-05-30 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer
Keywords: high dose radiotherapy; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
While surgery remains the standard treatment for rectal cancer, some patients still firmly refuse surgery for various reasons. Here, we conducted this retrospective observation study to discuss the feasibility of high-dose radiotherapy combined with chemotherapy in treating rectal cancer We retrospectively collect data of rectal cancer patients who were treated with high-dose radiotherapy plus chemotherapy in Sun Yat-sen University Cancer Center from April 1st, 2006 to July 30th, 2017. Patients gave up surgery before any treatment would have received one course of high dose radiotherapy (GTV60-70Gy/30-35f). Patients with tumor residual after neoadjuvant chemoradiotherapy but insisted non-operative treatment would have received 2 courses of radiotherapy (1st: GTV 45-50Gy/25f, 2nd: GTV 30/15f). The chemotherapy regimens included Capox, FOLFOX, or capecitabine at the discretion of the treating physician.

After treatment, patients were followed every 3 months for the first two years, at least every 6 months in the year thereafter. Recurrence, early and late toxicity were recorded.

Analyses were performed using SPSS software, version 19.0 (SPSS, Chicago, IL). Local recurrence and distant metastasis rate, progression free survival, and overall survival were calculated using the Kaplan Meier Method and were compared by log-rank test.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed diagnosis of rectal adenocarcinoma located within 15cm from the anal verge;
2. pelvic radiation with a total dose ≥60Gy for the treatment of rectal cancer;
3. refused surgery as the initial treatment;
4. a complete set of clinical information and follow-up data.

Exclusion Criteria:

1. patients with terminal cancer who received palliative treatment;
2. patients received any treatment before admission to Sun Yat-sen University Cancer Center;
3. patients with second primary cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included subjects identified from the database of the Sun Yat-sen University Cancer Center in the period of April 2006 to July 2017.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
clinical response rate | evaluate 5 weeks after radiotherapy
  the rate of clinical response in the whole group

SECONDARY OUTCOMES:
short term and long term side effects | from the complete to 3 years after treatment
  short term and long term toxicity related to high dose radiotherapy
progression free survival | 3 years
  defined as the time from the date of trial entry until disease progression, relapse, or death from any cause.
overall survival | 3 years
  calculated from the date of trial entry until death from any cause or was censored at last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China